CLINICAL TRIAL: NCT03286621
Title: Evaluation of Five Different Eye-tracking Paradigms to Determine Autism in Young Children
Brief Title: Development of Eye-tracking Based Markers for Autism in Young Children
Status: Completed | Type: Observational
Sponsor: University of Electronic Science and Technology of China (Other)
Responsible Party: Principal Investigator, Keith Kendrick, Professor, University of Electronic Science and Technology of China
Other Study IDs: UESCT_neuSCAN_41
Record Dates: First submitted 2017-09-14; First posted 2017-09-18 (Actual); Last update posted 2018-10-29 (Actual); Status verified 2018-10

CONDITIONS: Autism Spectrum Disorder
Keywords: eye tracking; visual preference
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Children with Autism Spectrum Disorder: Children with an Autism Spectrum Disorder according to DSM-5 criteria
  Interventions: Other: Administration of five eye-tracking paradigms
- Typically Developing Children: Typically developing children
  Interventions: Other: Administration of five eye-tracking paradigms
- Children with Delayed Development Disorders: Children with Delayed Developmental Disorders other than ASD
  Interventions: Other: Administration of five eye-tracking paradigms

INTERVENTIONS:
Other: Administration of five eye-tracking paradigms — All subjects will undergo the battery of five eye-tracking paradigms to determine potential markers for autism.

SUMMARY:
The main aim of the present study is to examine eye-tracking based markers for social processing deficits in children with autism spectrum disorder (ASD). To this end a battery of five eye-tracking paradigms will be administered to young children with ASD and typically developing children. To additionally evaluate the specificity of the eye-tracking markers a group of children with disorders of delayed development other than ASD will be included.

DETAILED DESCRIPTION:
During an initial screening session all participants will undergo the Autism Diagnostic Observation Schedule (ADOS). ASD-related symptomatology and levels of impairments will be further characterized using the Social Responsibilities Scale 2 (SRS 2), Caregiver Strain Questionnaire (CSQ), Aberrant Behavior Checklist (ABC), Social Communication Questionnaire (SCQ), and Repetitive Behaviour Scale Revised (RBS-R).

Subsequently all participants will be administered the following eye-tracking paradigms: (1) dynamic social and non-social visual preference paradigm during which dynamic geometric images (DGI) and dynamic social images (DSI) will be presented, (2) non-biological versus biological motion paradigm, (3) social attention and sharing of enjoyment paradigm, (4) preference for real versus schematic emotional face stimuli paradigm during which photographs of human faces and emoticons will be presented, (5) shared social attention and gaze direction paradigm.

ELIGIBILITY:
Exclusion criteria for all participants:

* visual, auditory or motor impairments
* use of medication

Inclusion criteria for all participants:

* written informed consent from parents / caregiver
* age: 1-10 years

Additional inclusion criterion for the ASD group:

- diagnosis of Autism Spectrum Disorder according to DSM-5

Additional inclusion criteria for typically developing children in the control group:

* no symptoms of developmental disorders
* no current or history of psychological disorder

Additional inclusion criterion for the unspecific disorder of delayed development children in the additional control group:

- disorder of delayed development other than ASD

Ages: 12 Months to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children with ASD according to DSM-5 criteria will be compared with typically developing children and a group of children with unspecific delayed development disorders.
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2017-09-09 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2018-02-28 (Actual)

PRIMARY OUTCOMES:
Global eye-gaze characteristics | Single assessment, total duration 20 minutes
  Global eye-gaze patterns between the three groups will be compared to determine ASD specific alterations
Feature-specific eye-gaze characteristics | Single assessment, total duration 20 minutes
  Localized feature-specific eye-gaze patterns will be compared between the three groups to determine ASD specific alterations

SECONDARY OUTCOMES:
Global eye-gaze characteristics and associations with symptom severity | Single assessment, total duration 20 minutes
  Associations between global eye-gaze characteristics and severity of ASD symptoms
Feature-specific eye-gaze characteristics and associations with symptom severity | Single assessment, total duration 20 minutes
  Associations between localized feature-specific eye-gaze patterns and severity of ASD symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Juan Kou, MSc, Study Chair — University of Electronic Science and Technology of China
Locations (1):
- School of Life Science and Technology, University of Electronic Science and Technology of China, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kou J, Le J, Fu M, Lan C, Chen Z, Li Q, Zhao W, Xu L, Becker B, Kendrick KM. Comparison of three different eye-tracking tasks for distinguishing autistic from typically developing children and autistic symptom severity. Autism Res. 2019 Oct;12(10):1529-1540. doi: 10.1002/aur.2174. Epub 2019 Aug 1. PMID 31369217